CLINICAL TRIAL: NCT05191628
Title: Amniotic Membrane Visio-AMTRIX in Recurrent Macular Hole
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual rate
Sponsor: TBF Genie Tissulaire (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Visio-AMTRIX-TMA-TBF; 2019-A01374-53 (Registry Identifier: IDRCB)
Record Dates: First submitted 2021-12-29; First posted 2022-01-13 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Macular Holes; Retinal Detachment
MeSH Terms: conditions — Retinal Perforations; Retinal Detachment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Visio-AMTRIX (Experimental): Disk of amniotic membrane apposed or buried on recurrent macular hole by the Investigator after vitrectomy and fluid-gas exchange.
  Interventions: Biological: Visio-AMTRIX

INTERVENTIONS:
Biological: Visio-AMTRIX — Chemically-treated, viro-inactivated, freeze-dried and irradiated amniotic membrane placed by the investigator during macular hole surgery

SUMMARY:
The purpose of this open, multicenter trial is to assess the impact of the use of an amniotic membrane graft on the closure of macular hole-associated retinal detachment in patients with failed previous macular surgery.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman over 18 years of age, less than 75 years
* Macular Hole of all etiologies
* Patient with history of opened macular hole after previous pars plana vitrectomy
* Delay between previous surgery and inclusion (relapse or non-closing hole) > 1 month
* Patient who received the study information and provided consent
* Patient who is a members or a beneficiary of a national health insurance plan

Exclusion Criteria:

* Ocular surgery other than the macular hole surgery in the prior 3 months
* Participation in other clinical studies in the prior 3 months
* Any current or prior ocular pathology that could interfere with the conduct of the study, including visually significant cataract or media opacity
* Patient with uncontrolled glaucoma on more than 1 intraocular lowering medication
* Patient with uveitis or other active ocular inflammation or infection
* Pregnant or breast-feeding woman. Women of childbearing age will be asked to undergo a pregnancy test before being enrolled into the study or to use an effective birth control method
* Person deprived of liberty by judicial or administrative measures
* Any other reason which in the opinion of the investigator would preclude the adherence of the schedules visits, safe participation in the study or affect the results of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Closure of recurrent macular hole | 6 months
  Macular hole closure evaluated by optical coherence tomography (OCT)

SECONDARY OUTCOMES:
Absence of adverse reaction | 7 days, 15 days, 1 month, 3 months, 6 months
  Analysis of all adverse events and comparison with adverse events observed after vitrectomy
Functional restoration after closure of the macular hole | 7 days, 15 days, 1 month, 3 months, 6 months
  Best corrected visual acuity (BCVA) and microperimetry assessment
Anatomical restoration | 1 month, 3 months, 6 months
  Anatomical restoration of the outer segments (external limiting membrane and ellipsoid layer). Anatomical changes in the ganglion cell layer of the retina in the area around the hole and under the membrane. The assessment is done by OCT measuring the thickness of the ganglion cell layer
Evaluation of the surgical technique of placing the membrane | 7 days, 15 days, 1 month, 3 months, 6 months
  Duration of coverage by Visio-AMTRIX and persistent after gas removal

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital de la Croix-Rousse, Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No